CLINICAL TRIAL: NCT06741163
Title: Effect of a Supplement Containing Olive Leaf Extract and Vitamins on Performance of Male Elite Cyclists
Acronym: NutriRide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: UCAM university (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2414NR
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Supplement; Endurance Cycling Performance; Endurance Exercise; Performance
Keywords: performance; cycling; supplement; endurance; oleuropein

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, two-arm parallel group study conducted in one center.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will be randomly allocated to receive the placebo, which is a water-based shot with similar appearance and taste but without the active ingredients of the test product. The placebo will be provided in sterilized Nalgene bottles of 60 mL, equivalent to one dose. Participants will consume one dose of the placebo before their training session on each intervention day (Day 5, Day 6, and Day 7).
  Interventions: Dietary Supplement: Placebo
- Intervention (Experimental): Participants will be randomly allocated to receive the test product, which is a water-based shot containing olive leaf extract (100mg Oleuropein), vitamins, and other active ingredients. The product will be provided in sterilized Nalgene bottles of 60 mL, equivalent to one dose. Participants will consume one dose of the test product before their training session on each intervention day (Day 5, Day 6, and Day 7).
  Interventions: Dietary Supplement: Pre-activity shot

INTERVENTIONS:
Dietary Supplement: Pre-activity shot — Water-based shot containing olive leaf extract (100mg Oleuropein), vitamins, and other active ingredients. The product will be provided in sterilized Nalgene bottles of 60 mL, equivalent to one dose. Participants will consume one dose of the test product before their training session on each intervention day (Day 5, Day 6, and Day 7).
  Arms: Intervention
Dietary Supplement: Placebo — Water-based shot with similar appearance and taste but without the active ingredients of the test product. The placebo will be provided in sterilized Nalgene bottles of 60 mL, equivalent to one dose. Participants will consume one dose of the placebo before their training session on each intervention day (Day 5, Day 6, and Day 7).
  Arms: Placebo

SUMMARY:
The study focuses on olive leaf extract, particularly its active component, Oleuropein, which has shown promise in enhancing energy metabolism and muscle performance in previous studies. Despite the existing evidence on the individual effects of olive leaf extract and various vitamins, there is a lack of data on their combined effects, especially in elite athletes. Therefore, the study aims to assess whether this supplement can positively influence perceived endurance, performance, mood, vitality, and fatigue during intensive training.

The study is a randomized, double-blind, placebo-controlled trial involving up to 40 male professional cyclists aged 21 to 36 years. Participants will be randomly assigned to either the test group, receiving the supplement, or the placebo group. The study will unfold over a 10-day period, including a baseline phase without the supplement and an intervention phase where participants will consume the product before training sessions.

The primary objective is to demonstrate that the supplement positively affects perceived endurance compared to a placebo. The primary endpoint will measure differences in average perceived endurance over three days of intense training. Secondary objectives include evaluating the effects of the supplement on perceived performance, mood, alertness, and physiological metrics (heart rate, power, cadence, and speed).

Participants will fill out questionnaires to assess their perceived endurance, performance, and mood before and after training sessions. Data on physiological performance will be collected through devices monitoring heart rate and other metrics. The study will employ mixed generalized linear regression models for statistical analysis, with a focus on superiority testing.

The study poses minimal risk to participants, as the investigational products have been previously tested for safety. No direct health benefits are anticipated from participation, but the research may contribute valuable insights into athletic performance enhancement.

Data collected will be securely managed and anonymized, adhering to Good Clinical Practices (GCP) and local regulations. Participants will be informed about the study's procedures and will provide informed consent prior to enrollment.

In summary, the NutriRide study seeks to explore the potential benefits of a supplement containing olive leaf extract and vitamins on the performance of elite male cyclists, aiming to fill gaps in current research on dietary interventions in sports performance.

DETAILED DESCRIPTION:
Olive leaf extract, particularly its active component Oleuropein, is of particular interest to the investigators due to the findings of a pre-clinical study, which demonstrated that this natural bioactive compound from olive leaf extract (OLE) enhanced energy metabolism, improved muscle performance, and reversed muscle decline. Furthermore, the clinical efficacy of OLE in supporting muscle energy metabolism has been validated in healthy adults. Other nutrients, such as B vitamins and guarana seed extract, have also been identified as essential for mitochondrial function and energy metabolism, improving attention, memory, mood, and alertness, particularly after intense exercise.

This study aims to build on these findings by administering a to professional cyclists a supplement rich in olive leaf extract, vitamins, and guarana seed extracts during their training camp and assessing its impact on their perceived endurance and performance.

The rationale for this project is grounded in the lack of available data on the combined effects of compounds such as OLE, B vitamins, magnesium and guarana extract, despite previous literature describing their individual effects on energy. The selection of professional cyclists as the study population is based on their high level of fitness and the rigorous physical demands they face during training. This makes them an ideal group for evaluating the potential benefits of the product on endurance and performance, and for generating new evidence on the potential advantages of such supplementation during the training phase of athletes.

The study involves the administration of a product and a placebo, both of which are water-based shots containing. Potential risks include adverse reactions to the product, although the ingredients have been tested in previous studies and found to be safe. Participants may experience discomfort from filling out the questionnaire 12 times in total.There are no direct health benefits expected for participants. The study aims to contribute to the scientific understanding of the effects of olive leaf extract on endurance and performance, which could benefit the wider athletic community. The study is considered to be of minimal risk due to the non-invasive nature of the procedures and the established safety profile of the investigational products.

The primary objective is to evaluate the superiority of the product supplemented with olive leaf extract and vitamins over the placebo in improving average perceived endurance after 3 days of intense exercise training. The secondary objectives of the study are to evaluate the effects of the supplement compared to placebo and baseline on:

1. Perceived performance during intense physical activity.
2. Subjective measures of mood and alertness after intense physical activity and their recovery overnight.
3. Heart rate, power, cadence, and speed during intense physical activity.

The study is a randomized, double-blind, placebo-controlled, two-arm parallel group study conducted in one center. The study design is adapted to follow the schedule of a 7-day training camp for professional cyclist organized in Moraira, Spain. The camp is composed of two training phases of 3 days with one day of rest in between. Participants in a study will be randomly assigned to either the test arm or the placebo arm at Day 0. During the first training phase of the camp, no participants will consume the test product or the placebo, and participants will answer questionnaires before and after each training session to assess their perception of endurance, performance, mood, and alertness. The participants heart rate, power, cadence, and speed will be monitored during training using various devices. In the second training phase, participants will consume the assigned products: the test arm will receive a supplement containing olive leaf extracts and vitamins before each training session, while the placebo group will receive a placebo shot. Each participant will consume 3 doses of either the test product or placebo, one for each training day.

The study will enrol up to 40 athletes from the TUDOR cycling team. The primary endpoint will be evaluated in the Full Analysis Set (FAS) following the intention-to-treat principle. The study will test the superiority of the product with a type I error set at 5%.

Participants will be randomly assigned to receive either the placebo or the product in a 1:1 ratio using block randomization. The analysis populations include the Intention-to-Treat (ITT), Safety Analysis Set (SAF), Full Analysis Set (FAS), and Per Protocol (PP).

Mixed generalized linear regression models will be used for data analysis. The primary endpoint will be tested in the FAS population using the least square mean estimated difference between groups. Superiority will be concluded if the 95% confidence interval lower boundary is above 0.

Study procedures: At the commencement of the training camp, participants will receive information about the study and will be invited to express their interest in participating.

Visit 0 (V0): During this initial visit, participants will meet with the team doctor or their representative to review the study procedures. Any questions will be addressed, and if the participant chooses to proceed, they will sign two original consent forms. One signed copy will be provided to the participant, while the second original copy will be retained by the study team. The team doctor will conduct an assessment to ensure that the participant meets the study criteria and will assign them to receive either the test product or the placebo. Participants will also be guided on how to download the app required to complete the necessary questionnaires directly on their phone. In order to conduct our study analyses, in addition to the data collected through the paper study questionnaires, data collected from various devices during the training camp, such as heart rate, power, cadence, and speed, will be utilized for study analyses. Participants will not need to take any additional actions regarding this data, as it will be obtained directly from their coach at the end of the training camp.

Visit 1 (V1): During this visit, the team doctor or a member of the study team will provide guidance on completing the necessary questionnaires related to self-perceived mood, alertness, performance, and fatigue. These parameters will be evaluated using a visual analogue scale, where participants will indicate the extent to which the described state applies to them at that moment.

Baseline Period (Day 1 - Day 3): Participants will be required to complete questionnaires before and after their longest training session each day from Day 1 to Day 3. Each session will take approximately 5 minutes.

Intervention Period (Day 5 - Day 7): In addition to filling out the questionnaires before and after the longest training session of the day, participants will be asked to consume the entire product provided on the day and confirm that they have taken it at the end of the day.

Follow-Up Period (24h after Day 7): After the last day of the intervention period, participants will be asked to report any adverse events occurring up to 24 hours after the last product intake to the team doctor in charge of the camp or their assistant. This can be done directly by phone.

Data will be entered from paper source documents into electronic Case Report Forms (eCRF). Participants will enter questionnaire data directly into the questionnaires paper form. Designated site personnel will have personal usernames and passwords to access the eCRF database, ensuring data security. All data modifications will be documented in an audit trail file, and the system complies with Good Clinical Practices (GCP) and e-signature laws.

Data will be collected from investigator site data, participant-reported outcomes, and external data sources (e.g., heart rate monitors, bike computers). The data manager will validate all data entered into the eCRF using automatic and manual queries to address discrepancies. Participant data will be anonymized and securely stored, with data transfer maintaining high standards of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males aged 21-36 years, inclusive, at enrolment.
2. Able to understand and to sign a written informed consent prior to study enrolment.
3. Willing and able to comply with the requirements for participation in this study.

Exclusion Criteria:

1. Currently participating in another interventional research study.
2. Family or hierarchical relationships with the research team members.
3. Any known/suspected food allergies. As reported by participant.

Ages: 21 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scales for self reported performance over 3 days of intense exercise training between the test group and the placebo group | From Day 5 to Day 7 (included)
  The difference in average perceived endurance will be assessed through Visual Analogue Scales over 3 days of intense exercise training between the test group that received a product supplemented with olive leaf extract and vitamins and the placebo group

SECONDARY OUTCOMES:
Visual Analogue Scales (VAS) on the difference in average perceived performance between the test group and the placebo group | Day 5 to Day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared to placebo on perceived performance, during intense physical activity, will be assessed through Visual Analogue Scales (VAS), over 3 days of intense exercise training between the test group and the placebo group.
Bond-Lader Visual Analogue Scales (BL-VAS) © on subjective measures of mood and alertness after intense physical activity and their recovery overnight | Day 5 to Day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared to placebo on subjective measures of mood and alertness after intense physical activity and their recovery overnight will be assessed through Bond-Lader Visual Analogue Scales (BL-VAS) © after physical activity and for the recovery overnight, over 3 days of intense exercise training of between the test group and the placebo group.
Difference in average heart rate, power, cadence & speed, over 3 days of intense exercise training between the test group and the placebo group. | Day 5 to Day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared to placebo on heart rate, power, cadence and speed during intense physical activity, will be measured thorugh the difference in average heart rate (Wahoo Trackr Heart Rate Monitor Chest Strap), power (SRAM Red AXS Quarrq power meter), cadence & speed (Wahoo Bolt V2 Bike computer), over 3 days of intense exercise training between the test group and the placebo group.
Visual Analogue Scales (VAS) on average perceived endurance and performance, over 3 days of intense exercise training between the baseline and the intervention periods. | Day 1 to day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared with baseline period on perceived endurance and performance, during intense physical activity, will be assessed by measuring difference in average perceived endurance and performance through a VAS questionnaire, over 3 days of intense exercise training between the baseline and the intervention periods.
Bond-Lader Visual Analogue Scales (BL-VAS) © on average mood and alertness after intense physical activity and their recovery overnight | Day 1 to day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared with baseline period on subjective measures of mood and alertness after intense physical activity and their recovery overnight will be assessed through BL-VAS©, over 3 days of intense exercise training of between the baseline and the intervention periods.
Difference in average heart rate (Wahoo Trackr Heart Rate Monitor Chest Strap), power (SRAM Red AXS Quarrq power meter), cadence & speed (Wahoo Bolt V2 Bike computer), between the baseline and the intervention per | Day 1 to day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared with baseline period on heart rate, power, cadence and speed during intense physical activity will be measured through the difference in average heart rate (Wahoo Trackr Heart Rate Monitor Chest Strap), power (SRAM Red AXS Quarrq power meter), cadence & speed (Wahoo Bolt V2 Bike computer), over 3 days of intense exercise training between the baseline and the intervention periods.
Visual Analogue Scales (VAS) on perceived endurance and performance during intense physical activity | Day 5 to Day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared to placebo, overtime, on perceived endurance and performance during intense physical activity will be assessed through a VAS questionnaire during 3 days of intense exercise training between the test group and the placebo group.
Difference in overtime heart rate, power, cadence & speed, over 3 days of intense exercise training between the test group and the placebo group. | Day 5 to Day 7 (included)
  The effect of consuming a supplement containing olive leaf extract and vitamins compared to placebo, overtime, on heart rate, power, cadence and speed during intense physical activity will be measured thorugh the difference overtime in heart rate (Wahoo Trackr Heart Rate Monitor Chest Strap), power (SRAM Red AXS Quarrq power meter), cadence & speed (Wahoo Bolt V2 Bike computer) during 3 days of intense exercise training between the test group and the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Serawa Moraira, Moraira, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared with the parties collaborating within this project:
  * UCAM
  * Tudor Cycling Professional Team
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD shared between November 2024 to May 2025
Access Criteria: The study PI and the Scientific Lead will be able to access the IPD through regulated virtual access to the electronic data capture (medidata) and trial master file (Veeva). To access all sensitive files, a software-specific and cloud-specific password and granted access will be required.
  If necessary, any transfer of files between the company and Nestlé will be conducted through their secure server, ensuring the confidentiality and security of the data.